CLINICAL TRIAL: NCT04000230
Title: Teacher-Child Interaction Training in Miami-Dade County Early Education Programs: A Randomized Control Trial
Brief Title: Teacher Child Interaction Training (TCIT): Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Children's Trust, Miami FL (Other)
Responsible Party: Principal Investigator, Eileen Davis, Assistant Professor of Clinical Pediatrics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20170372
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Behavior, Child
Keywords: Early Education Program; Developmental Delay; Behavior Management; Social Emotional Development; Special Education
MeSH Terms: conditions — Child Behavior; Learning Disabilities | interventions — Immunization, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCIT (Experimental): Teachers in the intervention group receive TCIT in the first half of the school year and booster coaching is provided throughout the second half of the school year as the Waitlist Control group is trained.
  Interventions: Behavioral: TCIT; Behavioral: Booster
- Waitlist Control (Active Comparator): Waitlist Control teachers do not receive any intervention for the first half of the school year. They then receive the same TCIT training as the intervention group in the second half of the school year.
  Interventions: Behavioral: TCIT

INTERVENTIONS:
Behavioral: TCIT — TCIT consists of the following:
  * CDI Teach Session: Teachers will participate in two training workshops in Child-Directed Interaction (CDI) skills. Specifically, teachers will learn to use positive attention skills and active ignoring.
  * CDI Coaching: Teachers will receive 90 minutes of CDI coaching in the classroom once or twice weekly for 6 total coaching sessions over a period of 4-6 weeks. The coach will observe the class and coach the teacher live using a microphone and bug-in-the-ear device.
  * TDI Teach Session: Teachers will complete two training workshops in Teacher Directed Interaction (TDI) skills, which focus on increasing compliance and reducing disruptive behavior. Teachers will learn to present developmentally appropriate, direct, and clear instructions and consistent positive and negative consequences.
  * TDI Coaching: Teachers will receive six 90-minute TDI coaching sessions once or twice weekly for 4-6 weeks.
Behavioral: Booster — Teachers in the Intervention group will receive additional booster sessions during the second half of the school year. Booster sessions consist of coaching teachers in CDI and TDI skills. Teachers receive 4-8 booster sessions.
  Arms: TCIT

SUMMARY:
This study is being conducted to evaluate the effects of TCIT on child development, child behavior, and teacher use of skills in the classroom.

ELIGIBILITY:
Inclusion Criteria:

* UMTCIT will target classrooms of children ages 1-5 enrolled in four participating B-2 Early Education Programs in Miami-Dade County: Debbie School, Easterseals South Florida, Arc of South Florida, and Linda Ray Intervention Center. Participants will also include school staff (teachers, teaching assistants, physical therapists, occupational therapists, speech/language pathologists) and students.

Exclusion Criteria:

* Children will be excluded from the study if they are 6 years of age or older or younger than 12 months of age at the start of each wave of treatment.

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in teacher use of TCIT skills | Baseline to 8 months
  Teacher-Child Interaction Coding System (TCICS) in a behavioral coding system that allows trained observers to tally the occurrence of certain teacher behaviors. For CDI skills, if teachers use the skills at a frequency of 5 or more each, they have demonstrated proficiency. If they use the skills at a frequency of 7 or more each, they have demonstrated mastery. For TDI skills, percent correct follow-up of commands and questions at a rate of 50% demonstrates proficiency. Percent correct follow-up at a rate of 75% demonstrates mastery.
Student social-emotional functioning | 8 months
  The Devereux Early Childhood Assessment (DECA) identifies each domain as an area of strength (T-score >=60), an area of need (T-score <=40), or an area of typical functioning (T-score = 41-59). DECA t-scores range from 28 to 72 with higher scores indicating higher functioning.
Child prosocial behaviors | 8 months
  The Behavior Assessment System for Children, Third Edition - Student Observation System (BASC-3 SOS) is a behavioral observation coding system that allows for interval recording of a wide range of child positive and negative behaviors that may promote or impede learning and adjustment in the classroom.
  For the Adaptive Behaviors scale, there are 4 behaviors rated across 30 intervals, for a total possible score of 120 (range 0-120). Higher scores on the Adaptive Behaviors scale are indicative of higher functioning.
Child disruptive/maladaptive behaviors | 8 months
  The Behavior Assessment System for Children, Third Edition - Student Observation System (BASC-3 SOS) is a behavioral observation coding system that allows for interval recording of a wide range of child positive and negative behaviors that may promote or impede learning and adjustment in the classroom.
  The Problem Behaviors scale consists of 10 behaviors rated across 30 intervals, for a total possible score of 300 (range 0-300). Higher scores on the Problem Behaviors scale are indicative of poorer functioning.

SECONDARY OUTCOMES:
Child disruptive behaviors | 8 months
  The Sutter-Eyberg Student Behavior Inventory-Related (SESBI-R) is a teacher rating scale of disruptive behavior of children. It is a 38-item questionnaire with each item scored from 1 (never) to 7 (always) for a total scoring range of 38-266. The higher score indicates increased child's disruptive behavior in the classroom setting.
Child language development | 8 months
  Assess early language based on the MacArthur Communicative Development Inventories (CDI). It is comprised of an 89-word vocabulary checklist. The score is assessed in the amount of correct answers and measured in percentiles, from less than 1 to 100, depending on the child's age. Higher percentile scores indicate a higher vocabulary (i.e., more language) and lower percentile scores indicate a lower vocabulary (i.e., less language).

CONTACTS AND LOCATIONS:
Overall Officials: Eileen M Davis, PhD, Principal Investigator — University of Miami
Locations (4):
- United States (4):
  - Debbie School, Miami, Florida
  - EasterSeals South Florida, Miami, Florida
  - Linda Ray Intervention Center, Miami, Florida
  - Arc of South Florida, Miami, Florida

IPD SHARING:
Plan to Share IPD: No